CLINICAL TRIAL: NCT00379730
Title: A Randomized, Double-blind Study of Treatment With a Known Anti-inflammatory (Prednisolone) to Evaluate Novel Endpoints in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Prednisolone Novel Endpoint Study in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: RES106087
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: CT scan; breathing tests; lung function tests; biomarkers; prednisolone; IOS; COPD; clinical outcomes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Prednisolone

SUMMARY:
Prednisolone will be used as a model medication to identify new clinical outcomes for future evaluation of new therapies in short-term studies (up to 4 weeks) in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* An established clinical history of COPD
* Evidence of bronchitis
* Current or ex-smoker

Exclusion Criteria:

* COPD exacerbation requiring steroid and/or antibiotics in the last month
* Taking oral or inhaled steroids for more than 14 days in the last 6 months
* Unable to withhold salbutamol/albuterol for a 6 hour period
* History of alcohol, substance or drug abuse within the last year.
* Other significant medical condition e.g. diabetes
* Cancer that has not been in complete remission for at least 5 years
* As a result of the medical interview, physical examination or screening investigations, that the doctor considers the subject unfit for the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2006-03-21; Study Completion 2007-05-03 (Actual)

PRIMARY OUTCOMES:
lung function tests using a system called Impulse oscillometry (IOS). CT scans to measure the thickness of the tubes in the lungs Blood, sputum and breath samples to measure chemical products in the lungs and body that relate to COPD

SECONDARY OUTCOMES:
Traditional lung function tests & Symptom Questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Mendoza, Argentina
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- GSK Investigational Site, Wellington, New Zealand
- GSK Investigational Site, Mowbray, South Africa

REFERENCES:
- [Derived] Lomas DA, Silverman EK, Edwards LD, Locantore NW, Miller BE, Horstman DH, Tal-Singer R; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints study investigators. Serum surfactant protein D is steroid sensitive and associated with exacerbations of COPD. Eur Respir J. 2009 Jul;34(1):95-102. doi: 10.1183/09031936.00156508. Epub 2009 Jan 22. PMID 19164344